CLINICAL TRIAL: NCT05750316
Title: Effect of Consumption of Cowpea Leaves on Postprandial Blood Glucose in Healthy Black Adults: A Randomised Controlled Pilot Study
Brief Title: Impact of Consumption of Cowpea Leaves on Postprandial Blood Glucose in Black Adults, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Charlotte E Mills, Lecturer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 06/2023
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Black Ethnicity
Keywords: Black ethnicity; Blood Glucose; Leaves; Cowpea; Vegetable
MeSH Terms: interventions — Junctional Adhesion Molecule A

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze dried cowpea leaves mixed in jam (Experimental): 6g of freeze-dried cowpea leaves (equivalent to one portion of vegetables) mixed with apricot jam and spread on bread.
  Interventions: Other: Cowpea leaves mixed with Jam
- Jam with green food colour (Active Comparator): Apricot jam mixed with green colouring and spread on bread
  Interventions: Other: Jam mixed with green food colour

INTERVENTIONS:
Other: Cowpea leaves mixed with Jam — 6g of freeze-dried cowpea leaves, equivalent to 80g(a portion) of vegetables mixed with Jam and spread on bread
  Arms: Freeze dried cowpea leaves mixed in jam
Other: Jam mixed with green food colour — Jam with green food colouring spread on bread
  Arms: Jam with green food colour

SUMMARY:
Intake of foods high in carbohydrates causes a spike in glucose in the blood. Repeated high blood glucose spikes are associated with an increased risk of diabetes. People of black ethnicity have higher risk of diabetes. Vegetables may help in the regulation of blood glucose. Cowpea, also referred to as black-eyed peas (Vigna unguiculata) leaves, contain polyphenols and fibre that can help regulate blood glucose.

The study will be an acute, single-blind, randomised control trial with a cross-over design involving healthy black participants aged ≥18 years. This clinical trial aims to investigate if consuming cowpea leaves can reduce blood glucose spikes after consuming a meal high in carbohydrates. Participants will be randomised to consume either bread with jam containing freeze-dried cowpea leaves (active intervention) or jam without any freeze-dried powder (control group). Blood glucose will be monitored before the intervention and every 15 minutes after the intervention using a continuous glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* Participants from Black, Black British, Caribbean or African ethnic backgrounds,which includes: Caribbean, African, Any other Black, Black British, or Caribbean background
* Should be able to give informed consent
* Should be willing to provide GP's contact details

Exclusion Criteria:

* Pregnant or lactating mothers
* Special dietary requirements such as vegetarians and vegans
* Participants who are on a specialised diet such as a weight reduction diet
* Having any chronic illness or taking medication for chronic illness
* Participants whose blood results indicate illness
* Participants on mediation for hypertension or hyperlipidaemia
* Sportsmen or women or vigorous exercise for more than 5 times per week
* Alcohol (more than 14 units per week) or drug abusers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose measured by incremental area under the curve and area under the curve | At baseline (t=0 hours) and 15 minutes interval until (t=3 hours)
  Postprandial blood glucose measured by a continuous glucose monitor. The incremental area under curve and area under the curve will be used as a measure of the postprandial blood glucose

SECONDARY OUTCOMES:
Change in blood pressure | At baseline (t=0 hours) and every 30 minute until (t=3 hours)
  Systolic and diastolic blood pressure by blood pressure monitor
Microvascular blood flow | At baseline (t=0 hours) and (t=2.5 hours)
  Microvascular blood flow using Laser doppler Imaging with Iontophoresis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No